CLINICAL TRIAL: NCT00484055
Title: Local Application of Collagen-Gentamicin in Addition to Fixation of the Sternum With Extra Sternal Wires for Prevention of Sternal Wound Infection in Cardiac Surgery
Brief Title: Local Collagen-Gentamicin and Extra Fixation of the Sternum for Prevention of Sternal Wound Infection in Cardiac Surgery
Acronym: LOGIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Orjan Friberg, MD, PhD, Region Örebro County
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OFR02
Record Dates: First submitted 2007-06-06; First posted 2007-06-08 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Drug Resistance, Bacterial; Postoperative Wound Infection
Keywords: Antibiotic Prophylaxis
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Active Comparator): Use of local CollagenGentamicin and enhanced sternal fixation according to the Clinical routine introduced 4 years earlier as a result of a previous RCT on 2000 patients. In that sense these patients did not receive any intervention but just the standard treatment introduced 4 years earlier.
  The aim of the study was to PROSPECTIVELY include a defined number of patients to compare their complication rate with that from aControl Group of patients från a previous RCT to verify that the effect of the treatment was stable over time.
  As the study did not include any intervention compared to the present standard treatment at that time ethical approval was Exempt.
  Interventions: Drug: Local application of collagen-gentamicin; Procedure: Fixation of the sternotomy with more than six wires

INTERVENTIONS:
Drug: Local application of collagen-gentamicin — Application of 2 sponges (5 x 20 cm) of collagen-gentamicin between the sternal halves immediately before sternal closure
  Other Names: Collatamp-G
Procedure: Fixation of the sternotomy with more than six wires — At least 7 (or more) sternal fixation wires (preferaby put as separate single wires) used for fixation of the sternum at wound closure

SUMMARY:
The aim of the present study is to evaluate a new technique for prevention of sternal wound infection consisting of local application of collagen-gentamicin in addition to routine i.v. antibiotic prophylaxis.

The technique has been evaluated in a previous randomised study. The aim of the present study is to evaluate the technique after it has been introduced in clinical practise to monitor the bacterial antibiotic susceptibility and to verify that the suggested reduction in sternal wound infection still exits.

DETAILED DESCRIPTION:
A new technique for prevention of sternal wound infections after cardiac surgery is studied. Local application directly in the surgical wound of aminoglycoside antibiotics (gentamicin) bound to collagen reduced the incidence of wound infection with more than 50 % in a previous prospective randomised trial.

As the technique has been introduced in clinical practise two questions need to be monitored:

* Are there signs of change in the bacteria that cause the wound infections with a shift over time towards more gentamicin resistant agents?
* Is the effect of the prophylaxis still comparable to that which was seen in the previous study?

Furthermore, results from the previous study indicated that the effect of the local antibiotic was better when combined with an extra rigid sternal wound infection, defined as at least one extra steel wire for sternal fixation.

The study is conducted at those two Swedish cardiothoracic surgery centers where it was first studied. There are thus two objectives of the study: first to analyze the microbiologic findings of the sternal wound infections that occur, and secondly to monitor the incidence of sternal wound infection (especially deep infections) when the local collagen-gentamicin prophylaxis is used in daily routine in combination with a specific surgical technique for optimization of the strength of sternal fixation.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive cardiac surgery patients operated via median sternotomy

Exclusion Criteria:

* Existing inclusion of the patient in another study of treatment aimed at reducing postoperative SWI.
* Known allergy or other contraindication to gentamicin or bovine collagen.
* Pregnancy or breast feeding
* Treatment with aminoglycosides during the last week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1358 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The incidences of methicillin- and gentamicin resistant microbiological agents in sternal wound infections that develop in study patients | Within 2 months postoperatively

SECONDARY OUTCOMES:
The absolute incidence of all SWI and of superficial SWI within 2 months and the relative (the ratio) incidences of superficial vs deep SW | 2 months postoperatively
The total incidence of SWI that requires surgical revision of the wound | 2 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Örjan Friberg, MD, PhD, Principal Investigator — Dept of Cardiothoracic Surgery and Anestesiology, University Hospital Orebro, Sweden
Locations (2):
- Sweden (2):
  - University Hospital, Dept of Cardiothoracic Surgery, Linköping
  - Dept of Cardiothoracic Surgery, University Hospital, Örebro

REFERENCES:
- [Background] Friberg O, Svedjeholm R, Kallman J, Soderquist B. Incidence, microbiological findings, and clinical presentation of sternal wound infections after cardiac surgery with and without local gentamicin prophylaxis. Eur J Clin Microbiol Infect Dis. 2007 Feb;26(2):91-7. doi: 10.1007/s10096-006-0252-6. PMID 17211605
- [Background] Friberg O, Dahlin LG, Soderquist B, Kallman J, Svedjeholm R. Influence of more than six sternal fixation wires on the incidence of deep sternal wound infection. Thorac Cardiovasc Surg. 2006 Oct;54(7):468-73. doi: 10.1055/s-2006-924437. PMID 17089314
- [Background] Friberg O, Svedjeholm R, Soderquist B, Granfeldt H, Vikerfors T, Kallman J. Local gentamicin reduces sternal wound infections after cardiac surgery: a randomized controlled trial. Ann Thorac Surg. 2005 Jan;79(1):153-61; discussion 161-2. doi: 10.1016/j.athoracsur.2004.06.043. PMID 15620935
- [Derived] Friberg O, Dahlin LG, Kallman J, Kihlstrom E, Soderquist B, Svedjeholm R. Collagen-gentamicin implant for prevention of sternal wound infection; long-term follow-up of effectiveness. Interact Cardiovasc Thorac Surg. 2009 Sep;9(3):454-8. doi: 10.1510/icvts.2009.207514. Epub 2009 Jun 18. PMID 19541691